CLINICAL TRIAL: NCT00540722
Title: A Phase 2 Study of R-(-)-Gossypol (Ascenta's AT-101) in Recurrent Glioblastoma Multiforme
Brief Title: Gossypol in Treating Patients With Progressive or Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00018; 0702; CDR0000569405; ABTC-0702; NABTT 0702; U01CA062475 (NIH)
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-07

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — gossypol acetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (R-(-)-gossypol acetic acid) (Experimental): Patients receive oral R-(-)-gossypol once daily on days 1-21. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Patients undergo tumor tissue and blood sample collection at baseline and periodically during study for biomarker correlative studies. Archived tumor tissue samples, if available, are analyzed for Bcl-2 family protein expression (e.g., Bcl-2, Bcl-xL, MCl-1, Bax, Bak, and BH3 domain for BH3 members only) and MGMT gene methylation status. Blood samples are analyzed for apoptotic protein levels (Bcl-2) by enzyme-linked immunosorbent assay.
  Interventions: Drug: R-(-)-gossypol acetic acid; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: R-(-)-gossypol acetic acid — Given PO
  Other Names: AT-101
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well gossypol works in treating patients with progressive or recurrent glioblastoma multiforme. Gossypol may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the overall survival rate associated with AT-101 in treating adult patients with recurrent glioblastoma multiforme.

SECONDARY OBJECTIVES:

I. To assess and estimate the acute and late toxicities. II. Tumor response rate. III. To estimate 6-month progression free survival. IV. To explore associations of the clinical outcome (overall survival) among the changes of potential serum biomarkers, baseline tumor protein expression and gene methylation status.

OUTLINE: This is a multicenter study.

Patients receive oral R-(-)-gossypol once daily on days 1-21. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo tumor tissue and blood sample collection at baseline and periodically during study for biomarker correlative studies. Archived tumor tissue samples, if available, are analyzed for Bcl-2 family protein expression (e.g., Bcl-2, Bcl-xL, MCl-1, Bax, Bak, and BH3 domain for BH3 members only) and 06-methylguanine-DNA-methyltransferase (MGMT) gene methylation status. Blood samples are analyzed for apoptotic protein levels (Bcl-2) by enzyme-linked immunosorbent assay.

After completion of study therapy, patients are followed every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed supratentorial glioblastoma multiforme which is progressive or recurrent after radiation therapy ± chemotherapy; patients with previously low grade glioma who progressed after radiotherapy ± chemotherapy and are biopsied and found to have glioblastoma multiforme are eligible
* Patients must have tumor tissue form completed and signed by a pathologist
* Patients must have measurable contrast enhancing progressive or recurrent glioblastoma multiforme by MRI or CT imaging (Within 14 days before starting treatment)
* Patients must have recovered from toxicity of prior therapy; an interval of at least 3 months must have elapsed since the completion of the most recent course of radiation therapy, while at least 3 weeks must have elapsed since the completion of a non-nitrosourea containing chemotherapy regimen, and at least 6 weeks since the completion of a nitrosourea containing chemotherapy regimen; NOTE: For non-cytotoxic, FDA approved agents (i.e. celebrex, thalidomide, etc.) therapy could be started 2 weeks after discontinuing this agent provided the patient has fully recovered from all toxicity associated with the agent; for investigational, non-cytotoxic agents a minimum of 3 weeks must have elapsed before the patient will be eligible for this study
* Patients must have a Karnofsky performance status >= 60% (i.e. the patient must be able to care for himself/herself with occasional help from others)
* Absolute neutrophil count >= 1500/mm^3
* Platelets >= 100,000/mm^3
* Creatinine =< 1.5mg/dl
* Total Bilirubin =< 1.5mg/dl
* Transaminases =< 2.5 times above the upper limits of the institutional norm
* Patients must be able to provide written informed consent
* Women of childbearing potential must have a negative serum pregnancy test; the effects of AT-101 on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because Bcl-2 inhibitors have the potential to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation, and for at least one month following the last dose of AT-101; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients must have a Mini Mental State Exam score >= 15

Exclusion Criteria:

* Patients with serious concurrent infection or medical illness which would jeopardize the ability of the patient to receive the treatment outlined in this protocol with reasonable safety; (Examples of medical illnesses are [but not limited to] the following: uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements)
* Patients who are pregnant or breast-feeding
* Patients who have received more than two prior treatments
* Patients who have been previously treated with gossypol, or have allergies to gossypol
* Patients receiving concurrent therapy for their tumor (i.e. chemotherapeutics or investigational agents); concurrent steroid use is allowed
* Patients with a concurrent malignancy are ineligible unless they are patients with curatively treated carcinoma-in-situ or basal cell carcinoma of the skin; patients with a prior malignancy are ineligible unless they have been free of disease for >= five years
* Patients with ≥ Grade 2 sensory neuropathy based on the NCI CTCAE
* Patients who are taking iron supplements
* Patients with any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow pills are excluded
* Patients cannot be receiving cytochrome P450-inducing anticonvulsants (EIAEDs; e.g., phenytoin, carbamazepine, phenobarbital, primidone, oxcarbazepine)
* Patients with malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel are excluded; subjects with ulcerative colitis, inflammatory bowel disease, or a partial or complete small bowel obstruction are also excluded
* Eligibility of patients receiving any other medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of AT-101 will be determined following review of their case by the Principal Investigator
* Patients with symptomatic hypercalcemia that is > Grade 2 (according to CTCAE)
* Requirement for routine use of hematopoietic growth factors (including granulocyte colony stimulating factor, granulocyte macrophage colony stimulating factor, or interleukin-11) or platelet transfusions to maintain absolute neutrophil counts or platelets counts above the required thresholds for study entry
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with AT-101; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Fiveash, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Moffitt Cancer Center, Tampa, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled on this study from Jan 2008 through September 2008. Patients were enrolled in an outpatient setting at 9 oncology clinical sites
Groups:
- Treatment (R-(-)-Gossypol Acetic Acid): Patients receive oral R-(-)-gossypol once daily on days 1-21. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Patients undergo tumor tissue and blood sample collection at baseline and periodically during study for biomarker correlative studies. Archived tumor tissue samples, if available, are analyzed for Bcl-2 family protein expression (e.g., Bcl-2, Bcl-xL, MCl-1, Bax, Bak, and BH3 domain for BH3 members only) and o6-methylguanine-DNA-methyltransferase (MGMT) gene methylation status. Blood samples are analyzed for apoptotic protein levels (Bcl-2) by enzyme-linked immunosorbent assay.
  R-(-)-gossypol acetic acid: Given PO
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (R-(-)-Gossypol Acetic Acid)
Started | 56
Completed | 56
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (R-(-)-Gossypol Acetic Acid): Patients receive oral R-(-)-gossypol once daily on days 1-21. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Patients undergo tumor tissue and blood sample collection at baseline and periodically during study for biomarker correlative studies. Archived tumor tissue samples, if available, are analyzed for Bcl-2 family protein expression (e.g., Bcl-2, Bcl-xL, MCl-1, Bax, Bak, and BH3 domain for BH3 members only) and MGMT gene methylation status. Blood samples are analyzed for apoptotic protein levels (Bcl-2) by enzyme-linked immunosorbent assay.
  R-(-)-gossypol acetic acid: Given PO
  laboratory biomarker analysis: Correlative studies
Arm/Group | Treatment (R-(-)-Gossypol Acetic Acid)
Number analyzed (Participants) | 56
Age, Continuous [Median (Full Range); unit: years] | 59 [34 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 53
  More than one race | 0
  Unknown or Not Reported | 0
Karnofsky Performance Status (KPS) [Median (Full Range); unit: units on a scale] — Karnofsky Performance Status Scale Higher score better 100 - Normal; no complaints; no evidence of disease; 90 - Able to carry on normal activity; minor signs or symptoms of disease, 80 - Normal activity with effort; some signs or symptoms of disease; 70 - Cares for self; unable to carry on normal activity or to do active work; 60 - Requires occasional assistance, but is able to care for most of his personal needs
  units on a scale | 80 [70 to 100]
Histology [Count of Participants; unit: Participants]
  Glioblastoma | 54
  Gliosarcoma | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: The overall failure rate will be estimated along with 95% confidence intervals. A median time of survival will be estimated using standard methods.
Time Frame: 4.5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (R-(-)-Gossypol Acetic Acid)
Number analyzed (Participants) | 56
months | 5.9 [3.9 to 7.3]

2. Secondary Outcome: Percent of Patients With Grade 3 and 4 Adverse Events Related to Treatment
Description: The proportion of patients with serious or life threatening (grade 3 and 4) toxicities will be estimated using NCI CTCAE
Time Frame: 3 years
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (R-(-)-Gossypol Acetic Acid)
Number analyzed (Participants) | 56
percentage of participants
  Seizure | 2
  IIeus | 2
  Hypophosphatemia | 2
  fatigue | 4
  Elevated troponin | 2

3. Secondary Outcome: Tumor Response Rate
Description: Complete response Complete disappearance of all tumor on MRI scan, off all glucocorticoids with stable or improving neurological exam minimum of 4 wks Partial response Greater than or equal 50% reduction in tumor size on MRI, on sable or decreasing glucocorticoids with stable or improving neurological exam for a minimum of 4 wks.
  Progressive disease Progressive neurological abnormalities not explained by other causes or greater than 25% increase in size of tumor or if new lesion.
  Stable disease Clinical status and MRI does not qualify for complete response, partial response or progression
Time Frame: 3 years
Population: 5 patients were not evaluable for response
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (R-(-)-Gossypol Acetic Acid)
Number analyzed (Participants) | 56
Participants
  Complete Response | 0
  Partial Response | 1
  Stable Disease | 15
  Progression | 35
  not evaluable | 5

4. Secondary Outcome: Progression-free Survival Rate, Defined as Patient Who is Alive and Disease Progression Free at the Time of 26-week (6 Months) From First Day of the Treatment
Description: The probability of 6-month progression-free survival will be estimated using binomial distribution.
Time Frame: 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (R-(-)-Gossypol Acetic Acid)
Number analyzed (Participants) | 56
months | 1.87 [1.87 to 2.17]

5. Other Pre Specified Outcome: Explore Clinical Outcome (Overall Survival) With Changes of Potential Serum Biomarkers, Baseline Tumor Protein Expression and Gene Methylation Status
Description: Archived tumor tissue and 1 serum sample pre first dose and 1 sample anytime during week 2 of cycle 1
Time Frame: 1 month
Population: no data to report. Not enough archived tumor tissue and survival outcome did not warrant an analysis of the Pharmacokinetics (PK)
Arm/Group | Treatment (R-(-)-Gossypol Acetic Acid)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: start of first dose until at least 30 days post last dose. approximately 3 years
Arm/Group | Treatment (R-(-)-Gossypol Acetic Acid)
Serious Adverse Events (participants affected / at risk) | 6/56
Other Adverse Events (participants affected / at risk) | 28/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (R-(-)-Gossypol Acetic Acid) (N=56)
Seizure (Nervous system disorders) | 1 (1)
lleus (Gastrointestinal disorders) | 1 (1)
hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
fatigue (General disorders) | 2 (2)
cardiac disorder other (Cardiac disorders) | 1 (1) — elevated troponin
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (R-(-)-Gossypol Acetic Acid) (N=56)
vomiting (Gastrointestinal disorders) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4)
peripheral sensory neuropathy (Nervous system disorders) | 4 (4)
fatigue (General disorders) | 21 (21)
diarrhea (Gastrointestinal disorders) | 3 (3)
constipation (Gastrointestinal disorders) | 4 (4)
anorexia (Metabolism and nutrition disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less